CLINICAL TRIAL: NCT07273656
Title: Efficacy and Safety of Cryotherapy Followed by Tirbanibulin Ointment for Actinic Keratosis on the Scalp and Forehead
Acronym: TIRBACRYO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Almirall, SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2023_0127
Record Dates: First submitted 2025-09-23; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Keratosis; Actinic Keratoses
Keywords: Tirbanibulin; Cryotherapy; Squamus cell carcinoma; Skin carcinoma; Actinic Keratosis; Field cancerization
MeSH Terms: conditions — Keratosis; Keratosis, Actinic | interventions — Cryotherapy; tirbanibulin

STUDY DESIGN:
Intervention Model Description: One single group, each patient serving as their own control, with an intra-individual comparison of one hemiscalp with the contralateral hemiscalp
Who Masked: Participant, Investigator
Masking Description: One single group, each patient serving as their own control, with an intra-individual comparison of one hemiscalp with the contralateral hemiscalp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Cryotherapy + Tirbanibulin : Tirbanibulin ointment applied once daily for 5 days, repeated 3 times (every 4 months)
  Interventions: Drug: Cryotherapy + Tirbanibulin
- Control group (Placebo Comparator): Cryotherapy + placebo : Tirbanibulin ointment applied once daily for 5 days, repeated 3 times (every 4 months)
  Interventions: Drug: Cryotherapy + Tirbanibulin

INTERVENTIONS:
Drug: Cryotherapy + Tirbanibulin — Tirbanibulin ointment applied once daily for 5 days, repeated 3 times (every 4 months)
  Other Names: Cryotherapy + placebo

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of a combined approach of cryotherapy and tirbanibulin for the treatment of actinic keratosis of the scalp and forehead, repeated every 4 months. A higher rate of complete response is expected with this combination compared to cryotherapy alone, as well as a better response with repeated treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years old presenting with ≥ 8 typical actinic keratoses (AK), clinically visible or palpable, grade I or II, with at least 4 AK per hemiscalp,
* Participants who, in the investigator's judgment, are in good general condition (ECOG ≤ 2),
* The AK must be distributed in 2 non-overlapping areas, and of similar grades,
* Patient capable of understanding and adhering to the study visit schedule and other protocol requirements,
* Patient capable of understanding and voluntarily signing informed consent,
* Patient covered by social insurance,
* Patient willing to comply with all study procedures and duration,
* Women of childbearing potential must:

Have a negative pregnancy test at screening and during the treatment period,

Use an effective contraceptive method throughout the study participation. Menopausal women (absence of menstruation for at least one year without other medical cause) or surgically sterile women (tubal ligation, hysterectomy, or bilateral oophorectomy) may be enrolled.

Exclusion Criteria:

* Clinically atypical and/or rapidly evolving actinic keratoses (AK) in the treatment area, and grade 3 AK according to Olsen classification,
* A defined treatment area that would be:

  1. Located somewhere other than the scalp and/or forehead,
  2. Within 5 cm of a wound that is not fully healed or a lesion suspicious for carcinoma,
* Prior treatment with tirbanibulin,
* Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for actinic keratoses in the treatment area or within 2 cm around this area within 6 weeks prior to the screening visit,
* Use of the following therapies within 2 weeks prior to the screening visit:

  1. Therapeutic or cosmetic procedures (e.g., liquid nitrogen application, surgical excision, dermabrasion, medium or deep chemical peeling, laser resurfacing) in the treatment area or within 2 cm around the selected treatment area,
  2. Therapeutic products containing acids (e.g., salicylic acid, fruit acids), topical retinoids, or light peels in the treatment area or within 2 cm around the selected treatment area,
* Allergy to tirbanibulin or any of its components.
* Any condition causing a risk of poor compliance,
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to sign the consent form,
* Women of childbearing potential who refuse to use an effective contraceptive method,
* Pregnant women, women planning to become pregnant, and breastfeeding women,
* Persons deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete clearance of actinic keratosis | 8 months
  Complete clearance rate of actinic keratoses at 8 months. A complete response corresponds to the absence of clinically detectable actinic keratosis in the treated area.

SECONDARY OUTCOMES:
To determine the 12-month effectiveness of a combined approach using cryotherapy and tirbanibulin. | 12 months
  Complete Clearance of Actinic Keratosis at 12 months. A complete response corresponds to the absence of clinically detectable actinic keratosis in the treated area.
To evaluate the reduction in the number of actinic keratoses after 2 treatment cycles. | 8 months
  Partial clearance rate (75% reduction in the number of actinic keratoses) at 8 months.
To evaluate the reduction in the number of actinic keratoses after 3 treatment cycles. | 12 months
  Partial clearance rate (75% reduction in the number of actinic keratoses) at 12 months.
To evaluate the reduction in the need for cryotherapy with tirbanibulin. | 12 months
  Number of cryotherapy sessions performed over the entire follow-up period.
To describe the safety and tolerability by treated side at each follow-up visit. | 12 months
  Safety: Local skin reactions assessed throughout the study

IPD SHARING:
Plan to Share IPD: No